CLINICAL TRIAL: NCT00640484
Title: Evaluation of the Effect of 2 Weeks Treatment With CHF 4226 pMDI 2µg and 4µg, Given Once Daily in the Morning, on 24-Hour FEV1 in Patients With COPD
Brief Title: Confirmatory Dose Finding Study of 2 Dosages of CHF 4226 pMDI (Carmoterol) in Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Steven E. Linberg, PhD, Chiesi Pharmaceuticals Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CCD-0706-PR-0026
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — carmoterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): CHF 4226 (carmoterol) 2 μg once a day, in the morning
  Interventions: Drug: carmoterol (CHF 4226)
- B (Experimental): CHF 4226 (carmoterol) 4 μg once a day, in the morning
  Interventions: Drug: carmoterol (CHF 4226)
- C (Placebo Comparator): placebo once a day, in the morning
  Interventions: Drug: placebo
- D (Active Comparator): salmeterol 50 μg twice daily, in the morning and in the evening
  Interventions: Drug: salmeterol

INTERVENTIONS:
Drug: carmoterol (CHF 4226) — carmoterol (CHF 4226) 2 μg once a day, in the morning
  (1 puff of carmoterol 2 μg + 1 puff of placebo pMDI)
  Other Names: CHF 4226; TA2005
  Arms: A
Drug: carmoterol (CHF 4226) — carmoterol (CHF 4226) 4 μg once a day, in the morning
  (1 puff of carmoterol 2 µg + 1 puff of carmoterol 2µg)
  Other Names: CHF 4226; TA2005
  Arms: B
Drug: placebo — placebo once a day, in the morning
  (1 puff of placebo pMDI + 1 puff of placebo pMDI)
  Arms: C
Drug: salmeterol — Salmeterol 50 μg twice daily, in the morning and in the evening
  (1 blister of Serevent Diskus BID)
  Other Names: Serevent Diskus/Accuhaler
  Arms: D

SUMMARY:
The purpose of this study is to confirm the dose of CHF 4226 (carmoterol) that should be given once a day to patients with COPD in order for the effect to last for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Signed IRB approved Informed Consent form
* Male or non-pregnant female, 40 -75 years old, inclusive
* Current or past cigarette smoking history of at least 15 pack-years
* Clinical diagnosis of COPD in accordance with recommendations of the National Heart Lung and Blood Institute/World Health Organization (NHLBI/WHO) Global Initiative for Chronic Obstructive Lung Disease (GOLD)
* Patient meets following requirements after FEV1 albuterol reversibility test (i.e., 30 minutes after 200μg (metered dose) albuterol MDI):

  * FEV1/FVC < 70%
  * FEV1 is at least 0.9L
  * FEV1 30% - 80%, inclusive, of patient's predicted normal value; ∆FEV1 > 5% of pre-albuterol value
  * If ∆FEV1 < 5% of pre-albuterol value, requirement must be met after retesting during run-in period, at least 24 hours prior to Period 1/Visit 1.

Exclusion Criteria:

* History of asthma
* Blood eosinophil count > 500/microliters
* History of allergic rhinitis or atopy
* COPD exacerbation or lower respiratory tract infection within 8 weeks prior to screening, or during run-in period, that resulted in use of an antibiotic, or oral or parenteral corticosteroids
* Inhaled corticosteroid that has been initiated, or effective dose has been changed, within 4 weeks prior to screening or during run-in period
* Uncontrolled cardiovascular (e.g., uncontrolled hypertension), respiratory, hematologic, immunologic, renal, neurologic, hepatic, endocrine (e.g., uncontrolled diabetes mellitus) or other disease, or any condition that might, in Investigator's judgment, place patient at undue risk or potentially compromise study results or interpretation
* History of coronary artery disease, cerebrovascular disease, cardiac arrhythmias
* Lung cancer or history of lung cancer
* Active cancer or history of cancer with < 5 years disease free survival time (with or without evidence of local recurrence or metastases). Localized basal cell carcinoma (without metastases) of skin is acceptable.
* Serum potassium value ≤ 3.5 mEq/L or > 5.5mEq/L and/or fasting serum glucose value ≥ 140 mg/dL
* Abnormal QTcF interval value in Screening visit ECG test (i.e., > 450 msec in males or > 470 msec in females)
* Cor Pulmonale
* Long term oxygen therapy, i.e., > 16 hours/24-hour period, every day, unless patient resides at elevation > 4000ft
* Use of any of the following medications prior to Screening, without meeting specified minimum washout period:

  * Long acting anti-cholinergic agent (i.e., tiotropium): 7 days
  * Short acting anti-cholinergics: 8 hours
  * Fixed combinations of β2-agonists and inhaled corticosteroids: 48 hours
  * Fixed combinations of an anti-cholinergic and short acting β2-agonist: 8 hours
* Long-acting β2-agonists: 48 hours
* Short acting β2-agonists (other than those prescribed in the study): 6 hours
* Theophylline and other xanthines: 1 week
* Parenteral or oral corticosteroids: 1 month
* Patient has taken any non-permitted medication
* Patient has received live-attenuated virus vaccination within two weeks prior to screening or during run-in (inactivated Influenza vaccination is acceptable if given > 48 hours prior to Screening)
* Known intolerance/hypersensitivity to β2-adrenergic agonists, propellant gases/excipients
* Patient is pregnant or lactating female, or female at risk of pregnancy (i.e., not using adequate contraceptive method: surgical sterilization [e.g., bilateral tubal ligation], hormonal contraception [implantable, patch, oral], IUD, and double-barrier methods [any double combination of: male or female condom with spermicidal gel, diaphragm, sponge, cervical cap]).
* Patient is mentally or legally incapacitated
* Patient has participated in another investigational study within 30 days prior to screening
* Abuse of alcohol or other substances
* Patient does not maintain regular day/night, waking/sleeping cycles (e.g., night shift worker)
* Patient is potentially non-compliant or unable to perform required protocol outcome measurements

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
FEV1 AUC0-24 standardized by time | on Day 15 (after 14 days of dosing)

SECONDARY OUTCOMES:
FEV1(L) | 30 min, 1, 2 ,3, 4, 6, 10, 12, 14, 16, 22, 23, and 24 hrs post dose at Visit 2 at all treatment periods
blood pressure | at the beginning and end of each of the four 14-day treatment periods
heart rate | at the beginning and end of each of the four 14-day treatment periods
FEV1 percent change | 30 min, 1, 2 ,3, 4, 6, 10, 12, 14, 16, 22, 23, and 24 hrs post dose at Visit 2 at all treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Donald P. Tashkin, MD, Principal Investigator — University of California, Los Angeles; Steven E. Linberg, PhD, Study Director — Chiesi Farmaceutici S.p.A.
Locations (15):
- United States (15):
  - Horizon Clinical Research Associates, PLLC, Gilbert, Arizona
  - Pulmonary Associates, PA, Phoenix, Arizona
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - University Clinical Research - DeLand, LLC, DeLand, Florida
  - Pulmonary Medicine and Critical Care, Austell, Georgia
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - Commonwealth BioMedical Research, Madisonville, Kentucky
  - North Carolina Clinical Research, Raleigh, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Asthma Allergy Associates, Portland, Oregon
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Reichman Associates, Sugar Land, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Matera MG, Cazzola M. ultra-long-acting beta2-adrenoceptor agonists: an emerging therapeutic option for asthma and COPD? Drugs. 2007;67(4):503-15. doi: 10.2165/00003495-200767040-00002. PMID 17352511
- [Background] Cazzola M, Matera MG, Lotvall J. Ultra long-acting beta 2-agonists in development for asthma and chronic obstructive pulmonary disease. Expert Opin Investig Drugs. 2005 Jul;14(7):775-83. doi: 10.1517/13543784.14.7.775. PMID 16022567
- [Background] Kikkawa H, Isogaya M, Nagao T, Kurose H. The role of the seventh transmembrane region in high affinity binding of a beta 2-selective agonist TA-2005. Mol Pharmacol. 1998 Jan;53(1):128-34. doi: 10.1124/mol.53.1.128. PMID 9443940
- [Background] Rossoni G, Manfredi B, Razzetti R, Civelli M, Bongrani S, Berti F. Positive interaction of the beta2-agonist CHF 4226.01 with budesonide in the control of bronchoconstriction induced by acetaldehyde in the guinea-pigs. Br J Pharmacol. 2005 Feb;144(3):422-9. doi: 10.1038/sj.bjp.0706096. PMID 15655502
- [Background] Rossoni G, Manfredi B, Razzetti R, Civelli M, Berti F. Positive interaction of the novel beta2-agonist carmoterol and tiotropium bromide in the control of airway changes induced by different challenges in guinea-pigs. Pulm Pharmacol Ther. 2007;20(3):250-7. doi: 10.1016/j.pupt.2006.01.004. Epub 2006 Mar 14. PMID 16533614
- [Background] Voss HP, Shukrula S, Wu TS, Donnell D, Bast A. A functional beta-2 adrenoceptor-mediated chronotropic response in isolated guinea pig heart tissue: selectivity of the potent beta-2 adrenoceptor agonist TA 2005. J Pharmacol Exp Ther. 1994 Oct;271(1):386-9. PMID 7965739
- [Background] Kikkawa H, Kanno K, Ikezawa K. TA-2005, a novel, long-acting, and selective beta 2-adrenoceptor agonist: characterization of its in vivo bronchodilating action in guinea pigs and cats in comparison with other beta 2-agonists. Biol Pharm Bull. 1994 Aug;17(8):1047-52. doi: 10.1248/bpb.17.1047. PMID 7820105
- [Background] Voss HP, Donnell D, Bast A. Atypical molecular pharmacology of a new long-acting beta 2-adrenoceptor agonist, TA 2005. Eur J Pharmacol. 1992 Dec 1;227(4):403-9. doi: 10.1016/0922-4106(92)90158-r. PMID 1359974
- [Background] Kikkawa H, Naito K, Ikezawa K. Tracheal relaxing effects and beta 2-selectivity of TA-2005, a newly developed bronchodilating agent, in isolated guinea pig tissues. Jpn J Pharmacol. 1991 Oct;57(2):175-85. doi: 10.1254/jjp.57.175. PMID 1687479
- [Background] Spadari-Bartfisch RC, Santos IN, Vanderlei LC, Marcondes FK. Pharmacological evidence for beta2-adrenoceptor in right atria from stressed female rats. Can J Physiol Pharmacol. 1999 Jun;77(6):432-40. PMID 10537229
- [Background] Matsukawa M, Takeda K, Shima H, Tagawa K, Banno K, Sato T. Enzyme-linked immunosorbent assay for TA-2005-glucuronide in human plasma. J Pharm Biomed Anal. 1998 Jun;17(2):245-54. doi: 10.1016/s0731-7085(97)00186-6. PMID 9638577